CLINICAL TRIAL: NCT06802315
Title: A Phase II Study of Intensity Modulated Total Marrow Irradiation (IM-TMI) in Addition to Myeloablative Fludarabine/Busulfan and Post-Transplant Cyclophosphamide (PTCY) for Fully Human Leukocyte Antigen (HLA)-Matched and Partially-HLA Mismatched Allogeneic Transplantation Patients With High-Risk AML, CML, and MDS
Brief Title: Intensity Modulated Total Marrow Irradiation in Fully Human Leukocyte Antigen (HLA)-Matched and Partially-HLA Mismatched Allogeneic Transplantation Patients With High-Risk Acute Myeloid Leukemia (AML), Chronic Myeloid Leukemia (CML), and Myelodysplastic Syndrome (MDS)
Acronym: BMT-13
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Matias Sanchez, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0865
Record Dates: First submitted 2025-01-28; First posted 2025-01-31 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia, Relapsed, Adult; Acute Myeloid Leukemia Refractory; Chronic Myeloid Leukemia - Accelerated Phase; Myelodysplastic Syndromes
Keywords: Total Marrow Irradiation; Stem Cell Transplant; Allogenic Transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia, Myeloid, Accelerated Phase; Myelodysplastic Syndromes | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Regimen (Experimental): Days -5 through -2: Fludarabine 40 mg/m2 IVPB daily and Busulfan targeting AUC 4800μM/min daily Day -3 through -1: Intensity modulated total marrow irradiation (9Gy fractionated) Day 0: Infuse peripheral blood mobilized stem cells Days +3 and +4: Cyclophosphamide 50 mg/kg/day Day 5: Mycophenolate mofetil and Tacrolimus (dose adjustment dependent on trough level) Day 30: Follow up Day 60: Follow up Day 90: Follow up Day 180: Follow up
  1. year: Follow up
  2. year: Follow up
  Interventions: Radiation: Intensity modulated total marrow irradiation; Drug: Cyclophosphamide (CTX); Drug: Fludarabine (Fludara); Drug: Busulfan (conditioning for ALLO Transplant)

INTERVENTIONS:
Radiation: Intensity modulated total marrow irradiation — See "Treatment Regimen"
Drug: Cyclophosphamide (CTX) — This study will determine the safety of the combination of Total Marrow Irradiation (TMI) and Post-Transplant Cyclophosphamide using a myeloablative fludarabine and iv targeted busulfan (Flu/Bu4) conditioning regimen.
Drug: Fludarabine (Fludara) — chemotherapy conditioning
Drug: Busulfan (conditioning for ALLO Transplant) — chemotherapy conditioning

SUMMARY:
The study is a Phase II clinical trial. Patients will receive intensity-modulated total marrow irradiation (TMI) at a dose of 9 Gray (Gy) with standard myeloablative fludarabine intravenous (IV) and targeted busulfan (FluBu4) conditioning prior to allogeneic hematopoietic stem cell transplant (HSCT). Graft-versus-host disease (GVHD) prophylaxis will include Cyclophosphamide on Day +3 and +4, tacrolimus, and mycophenolate mofetil.

DETAILED DESCRIPTION:
Patients will receive the following conditioning regimen: fludarabine 40 mg/m2 IV piggyback daily, from day -5 (5 days before stem cell infusion) through Day -2, IV busulfan targeting a 4800 μM/min/ day, from day -5 through day -2. In addition to the above chemotherapy, all patients will receive TMI at a dose of 3Gy on days -3, -2, and -1. On day 0, the stem cell product will be infused according to BMT (Bone Marrow Transplant) unit policy. Graft versus host disease (GVHD) prophylaxis will consist of the administration of Cyclophosphamide 50 mg/Kg on days 3 and 4 and mycophenolate mofetil combined with tacrolimus. Post-transplant evaluation will be done per standard care with study data collected at days 30, 60, 90, 180, 365, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-65 years.
* 2. Patients with CML, AML, or MDS who meet one of the following criteria: 2a. Relapsed or refractory AML (including AML in CR2) 2b. Poor-risk AML in first remission, with remission defined as <5% bone marrow blasts morphologically:
* AML arising from MDS, a myeloproliferative disorder, or secondary AML
* Poor risk molecular features according to Leukemia Net including ASXL1, BCOR, EZH2, RUNX1, SF3B1, SRSF2, STAG2, U2AF1, and/or ZRSR2
* Poor-risk cytogenetics: Monosomal karyotype, complex karyotype (> 3 abnormalities), inv (3), t(3;3), t(6;9), MLL rearrangement with the exception of t(9;11), or abnormalities of chromosome 5 or 7. 2c. Primary refractory disease 2d. MDS with at least one of the following poor-risk features:
* Poor-risk cytogenetics including 3q abnormalities, 7/7q minus or complex cytogenetics (>3 abnormalities).
* Current or previous INT-2 or high IPSS score.
* Treatment-related MDS.
* MDS diagnosed before the age of 21 years.
* Progression on or lack of response to standard DNA-methyltransferase inhibitor therapy.
* Life-threatening cytopenias, including those requiring regular PRBC or platelet transfusions. 2e. CML with a history of accelerated or blast phase.

Exclusion Criteria:

* 1. Presence of significant co-morbidity as shown by:
* 1a. Left ventricular ejection fraction < 50%
* 2b. Creatinine clearance <30ml/min.
* 3c. Bilirubin > 2.0 mg/dL (unless due to Gilbert's syndrome or hemolysis), and ALT and AST > 5 x ULN.
* 4d. FEV1 and FVC < 50% of predicted or DLCO <50% of predicted once corrected for anemia.
* 5e. Karnofsky score <70
* 6f. Active viral hepatitis or HIV infection.
* 7g. Cirrhosis.
* 2. Pregnancy or breast feeding
* 3. Patients unable to sign informed consent.
* 4. Patients previously received radiation to >20% of bone marrow-containing areas.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
GVHD-Free Relapse-Free Survival after Stem Cell Transplant | 1 Year Post-Stem Cell Transplant
  The 1-year GVHD- free relapse-free survival after HSCT (hematopoietic stem cell transplantation) conditioned with a 9Gy TMI in combination with FluBu4 and PTCY in patients with acute myeloid leukemia (AML), chronic myeloid leukemia (CML), Myelodysplastic Syndrome (MDS) at high risk of relapse.

SECONDARY OUTCOMES:
Overall Survival | 2 Years Post-Stem Cell Transplant
  The number of participants who have overall survival
Time To Engraftment | 30 Days Post-Stem Cell Transplant
Adverse Events | 30 Days Post-Stem Cell Transplant
  The number of adverse events and grades of severity per Common Terminology of Criteria for Adverse Events (version 5.0) and the Bearman scale.
Adverse Events | 60 Days Post-Stem Cell Transplant
  The number of adverse events and grades of severity per Common Terminology of Criteria for Adverse Events (version 5.0).
Adverse Events | 90 Days Post-Stem Cell Transplant
  The number of adverse events and grades of severity per Common Terminology of Criteria for Adverse Events (version 5.0)
Adverse Events | 180 Days Post-Stem Cell Transplant
  The number of adverse events and grades of severity per Common Terminology of Criteria for Adverse Events (version 5.0).
Adverse Events | 1 Year Post-Stem Cell Transplant
  The number of adverse events and grades of severity per Common Terminology of Criteria for Adverse Events (version 5.0).
Incidence of Acute Graft Versus Host Disease | 30 Days Post-Stem Cell Transplant
  The number of participants with Acute Graft Versus Host Disease
Incidence of Acute Graft Versus Host Disease | 60 Days Post-Stem Cell Transplant
  The number of participants with Acute Graft Versus Host Disease
Incidence of Acute Graft Versus Host Disease | 90 Days Post-Stem Cell Transplant
  The number of participants with Acute Graft Versus Host Disease
Incidence of Acute Graft Versus Host Disease | 180 Days Post-Stem Cell Transplant
  The number of participants with Acute Graft Versus Host Disease
Incidence of Acute Graft Versus Host Disease | 1 Year Post-Stem Cell Transplant
  The number of participants with Acute Graft Versus Host Disease
Incidence of Chronic Graft Versus Host Disease | 180 Days Post-Stem Cell Transplant
  The number of participants with Chronic Graft Versus Host Disease
Incidence of Chronic Graft Versus Host Disease | 1 Year Post-Stem Cell Transplant
  The number of participants with Chronic Graft Versus Host Disease
Transplant-Related Mortality | 30 Days Post-Stem Cell Transplant
  The number of participants with transplant-related mortality
Transplant-Related Mortality | 60 Days Post-Stem Cell Transplant
  The number of participants with transplant-related mortality
Transplant-Related Mortality | 90 Days Post-Stem Cell Transplant
  The number of participants with transplant-related mortality
Transplant-Related Mortality | 180 Days Post-Stem Cell Transplant
  The number of participants with transplant-related mortality
Transplant-Related Mortality | 1 Year Post-Stem Cell Transplant
  The number of participants with transplant-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Matias Sanchez, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States